CLINICAL TRIAL: NCT02115828
Title: A Pharmacodynamic Study of Vismodegib in Men With Metastatic Castration-resistant Prostate Cancer (mCRPC) With Accessible Metastatic Lesions for Tumor Biopsy
Brief Title: A Study of Vismodegib in Men With Metastatic CRPC With Accessible Metastatic Lesions for Tumor Biopsy
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J1423; NA_00093427 (Other: JHMI-IRB)
Record Dates: First submitted 2014-04-14; First posted 2014-04-16 (Estimated); Results first posted 2018-07-20 (Actual); Last update posted 2018-07-20 (Actual); Status verified 2017-10

CONDITIONS: Prostate Cancer
Keywords: Vismodegib; Metastatic Castration-Resistant Prostate Cancer; Accessible Metastatic Lesions for Tumor Biopsy
MeSH Terms: conditions — Prostatic Neoplasms | interventions — HhAntag691

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Vismodegib (Experimental): Vismodegib Treatment arm will receive Vismodegib by mouth 150 mg daily up to 1 year.
  Interventions: Drug: Vismodegib

INTERVENTIONS:
Drug: Vismodegib

SUMMARY:
This is a single-arm pharmacodynamic study with mandatory metastatic tumor biopsies in men with castration-resistant prostate cancer.

The trial will evaluate the effect of vismodegib on tumor tissue in men with metastatic CRPC by obtaining tumor biopsies at baseline and after 4 weeks of treatment with vismodegib.

DETAILED DESCRIPTION:
The study will enroll 10 evaluable patients. Patients will receive a 30-day supply of 150 mg of vismodegib on day one of each cycle daily by mouth, beginning on Day 1, and continuously until one of the following occurs: Disease progression, intolerable toxicity most probably attributable to vismodegib or withdrawal from the study.

Tumor biopsies (nodal or visceral), skin biopsies, and CTCs will be obtained at baseline and after 4 weeks of treatment. PSA evaluations will be conducted every 4 weeks, imaging assessments (CT and Bone scan) will be conducted every 12 weeks and routine labs (blood counts and chemistry panel) will be conducted every 4 weeks.

The investigator's intent is to examine the fold change in GLI1 expression in each man following exposure to drug (comparing pre-treatment and on-treatment core biopsy samples). As secondary endpoints, the investigator will also explore clinical response (PSA responses, progression-free survival [PFS], radiographic responses), safety, and will examine changes from baseline in Gli2, PTCH1, and AKT1 mRNA levels by qRT-PCR, in situ GLI1 expression in tissue sections by mRNA in situ hybridization, and GLI1 expression in isolated circulating tumor cells (CTCs).

ELIGIBILITY:
Inclusion Criteria:

* Men with metastatic castration-resistant prostate cancer (mCRPC), with accessible metastatic soft-tissue lesions for tumor biopsy
* Greater than 18 years of age
* Evidence of disease progression (PSA progression, or radiographic/clinical progression [PCWG2])

  * PSA progression is defined as at least two consecutive rises in serum PSA, obtained at a minimum of 1-week intervals, and each value ≥ 2.0 ng/mL.
  * Radiographic progression is defined for soft tissue lesions using RECIST criteria, i.e. an increase greater than 20% in the sum of the longest diameter of all target lesions based on the smallest sum longest diameter since treatment started or the appearance of one of more new lesions with a confirmatory scan 6 or more weeks later. Radiographic progression will be defined for bone lesions as the appearance of two new lesions with a confirmatory scan performed 6 or more weeks later that shows at least 2 or more additional new lesions.
* Presence of ≥1 metastatic site (nodal, visceral) that is amenable to core biopsy
* Castrate serum testosterone (<50 ng/dL)
* Prior anti-androgens are permitted but not required (2 week washout from anti-androgens)
* Prior abiraterone and enzalutamide are permitted (2 week washout for both agents)
* Prior immunotherapy (e.g. sipuleucel-T), and chemotherapy are permitted (4 week washout period from chemotherapy)
* Bisphosphonates and denosumab are permitted, if on a stable dose for ≥4 weeks
* Life expectancy ≥12 months
* Adequate renal, liver, and bone marrow function with the following acceptable initial laboratory values:

  * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) must be ≤ 2.5 x the upper limit of normal (ULN).
  * Total bilirubin must be ≤ 1.5 x ULN.
  * Estimated creatinine clearance using the Cockcroft-Gault formula must be > 40 mL/minute (See section 12.2 for formula)
  * Absolute neutrophil count (ANC) must be ≥ 1500/μL
  * Platelet count must be ≥ 100,000/μL
* Willing and able to provide written informed consent and HIPAA authorization for the release of personal health information.

NOTE: HIPAA authorization may be either included in the informed consent or obtained separately.

* Karnofsky Performance status/ECOG Performance Status ≥70/2 (Appendix A: Performance Status Criteria)
* Male patients must use condoms at all times, even after a vasectomy, during sexual intercourse with female partners of reproductive potential during treatment with vismodegib and for 2 months after the last dose to avoid exposing a pregnant partner and unborn fetus to vismodegib.

Exclusion Criteria:

* Current use of systemic corticosteroids (>5 mg prednisone)
* Known brain metastases, or untreated meningeal/dural disease
* Receiving any other investigational agents or receipt of another investigational agent within 4 weeks of study entry
* Patients taking anticoagulants or with a history of a bleeding diathesis (due to need for visceral biopsy)
* Use of any prohibited concomitant medications (washout period of 1 week)
* Insufficient time from last prior regimen or radiation exposure (washout period of 4 weeks)
* Grade > 2 treatment-related toxicity from prior therapy
* Any other condition which, in the opinion of the Investigator, would preclude participation in this trial

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2014-04; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel Antonarakis, M.D., Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

REFERENCES:
- [Result] Maughan BL, Suzman DL, Luber B, Wang H, Glavaris S, Hughes R, Sullivan R, Harb R, Boudadi K, Paller C, Eisenberger M, Demarzo A, Ross A, Antonarakis ES. Pharmacodynamic study of the oral hedgehog pathway inhibitor, vismodegib, in patients with metastatic castration-resistant prostate cancer. Cancer Chemother Pharmacol. 2016 Dec;78(6):1297-1304. doi: 10.1007/s00280-016-3191-7. Epub 2016 Nov 8. PMID 27826729

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 9 patients were enrolled on the study
Groups:
- Vismodegib: Vismodegib Treatment arm will receive Vismodegib by mouth 150 mg daily up to 1 year.
  Vismodegib
Period: Overall Study
Arm/Group | Vismodegib
Started | 9
Completed | 9
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All patients were required to have biopsies of the tumor and skin (a surrogate tissue) at baseline and after 4 weeks of therapy. 9 patients were enrolled. A nuclear medicine bone scan and CT scan of the C/A/P were performed to establish a baseline of the metastatic disease burden.
Arm/Group | Vismodegib
Number analyzed (Participants) | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 0
Age, Continuous [Median (Full Range); unit: years] | 65 [58 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 9
Region of Enrollment [Number; unit: participants]
  United States | 9

OUTCOME MEASURES:

1. Primary Outcome: The Proportion of mCRPC Patients Treated With Vismodegib Who Achieve a Pharmacodynamic (PD) Response in Tumor Biopsies
Description: The primary endpoint is the proportion of mCRPC patients treated with vismodegib who achieve a pharmacodynamic (PD) response in tumor biopsies, defined as both a decrease in GLI1 mRNA greater than 1.2 times the standard deviation (SD) of the baseline values and a ≥50% (≥2-fold) reduction in GLI1 messenger ribonucleic acid (mRNA) expression in metastatic tumor biopsies after 4 weeks of treatment when comparing post-treatment biopsy to pre-treatment biopsy in the same patient.
Time Frame: Up to 1 year
Population: The design had 90% power to detect a true 65% PD response rate across patients, with a false-positive rate of 3.3% under the null hypothesis that vismodegib has no effect in downregulating Gli1 expression.
Measure: Count of Participants; unit: Participants
Arm/Group | Vismodegib
Number analyzed (Participants) | 9
Participants | 7

2. Secondary Outcome: GLI1 Expression
Description: Suppression by vismodegib in tumor tissue of Hh-regulated transcripts and proteins was defined as the change from baseline in expression levels of GLI1 in situ tissue expression by mRNA in situ hybridization.
Time Frame: Up to 1 Year
Population: One patient did not receive a post-treatment biopsy, and another patient had insufficient tissue for evaluation from the repeat biopsy
Measure: Median (Full Range); unit: expression fold change
Arm/Group | Vismodegib
Number analyzed (Participants) | 7
expression fold change | -9.8 [-8841 to 122]

3. Secondary Outcome: Progression-free Survival (PFS)
Description: Progression-free survival (PFS) is defined by the Prostate Cancer Working Group 2 (PCWG2) criteria using RECIST 1.1 criteria for each patient. PFS is defined as the time of first dose (a) until prostate specific antigen (PSA) progression (by 25% increase in PSA from nadir) or death and (b) until any evidence of progression (by 25% increase in PSA from nadir, a new lesion on bone or CT scan, or physical examination) or death. PFS will be assigned to the earliest observed time.
Time Frame: Up to 1 Year
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Vismodegib
Number analyzed (Participants) | 9
months | 1.9 [1.3 to 1.9]

4. Secondary Outcome: AKT1 Expression in Tumor Biopsies
Description: The tumor biopsies were evaluated for changes to Hh-regulated transcript, AKT1, between pre-treatment and post-treatment
Time Frame: Up to 1 Year
Population: as for outcome 2
Measure: Median (Full Range); unit: expression fold change
Arm/Group | Vismodegib
Number analyzed (Participants) | 7
expression fold change | -1.15 [-5.28 to 2.93]

5. Secondary Outcome: The Effect of Vismodegib on PSA Responses
Description: The effect of vismodegib on PSA responses will be assessed as the number of patients with participants with ≥50% PSA reductions at any time point during study
Time Frame: Up to 1 Year
Population: Seven patients were evaluable for PSA response. One participant had no measurable PSA production at enrollment, and PSA remained <0.01 throughout the study. A second patient had disease progression prior to the first on-study PSA evaluation.
Measure: Number; unit: participants
Arm/Group | Vismodegib
Number analyzed (Participants) | 7
participants | 1

ADVERSE EVENTS:
Arm/Group | Vismodegib
Serious Adverse Events (participants affected / at risk) | 5/9
Other Adverse Events (participants affected / at risk) | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vismodegib (N=9)
chest pain and shortness of breath (Cardiac disorders) | 1 (1) — This is a 65 yr old man with Prostate CA , admitted for chest pain and shortness of breath. A cardiac event was ruled out. The cause of his symptoms appeared to be related to his metastatic prostate cancer process.
observation post-TACE (Hepatobiliary disorders) | 1 (1) — 60 year old man with prostate cancer underwent TACE to his liver metastases and and was admitted to the hospital for one night for observation post-TACE. This hospitalization was NOT RELATED to the study drug, vismodegib
Pain grade 3 (General disorders) | 1 (1) — patient was admitted om 07/15/2015 for pain control issues, SAE was not related to the study drug
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) — patient was admitted for grade 3 pneumonia. the SAE was not related to the study drug
Nausea (Gastrointestinal disorders) | 1 (1) — Patient was admitted for grade 3 nausea, the SAE was possibly related to the study drug
vomiting (Gastrointestinal disorders) | 1 (1) — Patient was admitted for grade 3 vomiting, this SAE was possibly related to the study drug.
Dehydration (Metabolism and nutrition disorders) | 1 (1) — Patient was admitted for grade 3 dehydration, the SAE was possibly related to the study drug
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vismodegib (N=9)
dysgeusia (Nervous system disorders) | 3 (4)
anorexia (Metabolism and nutrition disorders) | 3 (5)
fatigue (General disorders) | 6 (9)
nausea (Gastrointestinal disorders) | 6 (6)
vomiting (Gastrointestinal disorders) | 4 (4)
musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 6 (12)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes